CLINICAL TRIAL: NCT01666639
Title: Behavioral Exercise Therapy to Optimize Inpatient Behavioral Orthopedic Rehabilitation for Chronic Non-specific Low Back Pain
Brief Title: Behavioral Exercise Therapy and Multidisciplinary Rehabilitation for Chronic Non-specific Low Back Pain
Acronym: VBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Deutsche Rentenversicherung (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Prof. Dr., University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0421-FSCP-Z256
Record Dates: First submitted 2012-06-18; First posted 2012-08-16 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Behavioral: Usual Behavioral Medical Rehabilitation
- Intervention Group (Experimental)
  Interventions: Behavioral: Behavioral Medical Rehabilitation plus behavioral exercise therapy

INTERVENTIONS:
Behavioral: Behavioral Medical Rehabilitation plus behavioral exercise therapy — The Intervention Group is characterized by the same treatment as in the control group, plus a modification of the exercise therapy. An "Behavioral Exercise Therapy" (BET) is implemented in the usual care. The Behavioral Exercise Therapy is based on a goal-oriented and systematic combination of knowledge-, behavior-, and exercise-related elements. It had been developed prior as part of a multidisciplinary treatment and was adapted for this study. The Aims of BET are gradual improvements of individual coping competencies and self-management regarding back pain as well as long-term adherence to physical activity.
  Arms: Intervention Group
Behavioral: Usual Behavioral Medical Rehabilitation — The Behavioral Medical Rehabilitation (BMR), which is in this case the control group (usual care), consists of usual orthopedic medical care, exercise therapy, individual physiotherapy, psychological treatment elements (e.g. a pain management group), occupational therapy and back school. Pain medication is given if necessary. For the most part, the psychological elements draw a distinction between more "traditional" concepts or orthopedic rehabilitation and the BMR. The pain management group with its cognitive-behavioral principles comprises 9 sessions of 90 minutes each.
  Arms: Control Group

SUMMARY:
Multidisciplinary behavioral-orthopedic rehabilitation in the treatment of chronic back pain has proven its short-term effectiveness. Exercise therapy plays a major role in such a combination of treatments. There is a considerable need to develop theory-based exercise interventions which foster a long-term adherence to physical activity. Furthermore, an integration of behavioral elements such as coping competencies regarding back pain is needed. It is not yet clear, which specific part of multidisciplinary rehabilitation causes its effects. The role of exercise therapy has yet to be investigated. Aim of this study is the implementation of a standardized behavioral exercise therapy into an existing behavioral-medical rehabilitation for patients with chronic back pain. The main hypothesis is that the participation in the behavioral exercise therapy leads to greater short- and long-term improvements in functional capacity compared to the usual care.

ELIGIBILITY:
Inclusion Criteria (ICD-10):

* F45.4 Persistent somatoform pain disorder
* F45.41 Chronic pain disorder with somatic and psychological factors
* F54 Psychological and behavioural factors associated with disorders or diseases classified elsewhere
* M51.2 Other specified intervertebral disc displacement
* M51.3 Other specified intervertebral disc degeneration
* M51.4 Schmorl's nodes
* M51.8 Other specified intervertebral disc disorders
* M51.9 Intervertebral disc disorder, unspecified
* M53.8 Other specified dorsopathies
* M53.9 dorsophathy, unspecified
* M54.4 Lumbago with sciatica
* M54.5 Low back pain
* M54.6 Pain in thoracic spine
* M54.8 Other dorsalgia
* M54.9 Dorsalgia, unspecified
* R52.2 Other chronic pain

Exclusion Criteria:

* distinct specific diagnosis for back pain (e.g. radicular symptoms, myelopathy)
* severely limited health status (comorbidity)
* serious impairment of vision and hearing (not corrected)
* serious psychiatric codiagnosis (exkl. see inclusion criteria)
* inability to speak german
* pension claim (§51 SGB V - german law)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Hannover Functional Ability Questionnaire (HFAQ) (Kohlmann, Raspe, 1996) | one year
  The Hannover Functional Ability Questionnaire surveys the subjective estimate of a person of his or her functional ability in the context of physical activities of daily living. The Questionnaire has 12 Items. The participant is asked whether he or she is able to perform activities (e.g. to put on and pull off one's socks) and rates each on a 3-point scale (1=yes, 2=yes, but with trouble), 3=no, or only with help).

SECONDARY OUTCOMES:
Freiburger Questionnaire on Physical Activity (FQPA) (Frey et al., 1999) | one year
  The FQPA measures the amount of physical activity in different contexts performed by the participants: occupational setting (rating: intensive movement, moderate movement, mostly sitting) as well as leisure time physical activity (e.g. gardening, stair-climbing, habitual walking and cycling, sports). It consists of eight items.
Numeric Rating Scale (NRS) to assess pain intensity (Farrar et al., 2001) | one year
  Three items to assess the pain intensity felt by participants at the moment, as well as during the last six months (mean and maximum pain).
Graded Chronic Pain Status (GCPS)(von Korff et al., 1992)(adapted for 6 months) | one year
  Six items to assess the number of days with pain during the last six months, the history of pain and the functional disability due to pain.
Generalized Anxiety Disorder (GAD-7) (Löwe et al., 2008) | one year
HAPA variables (Fleig et al., 2011; Sniehotta et al., 2005; Schwarzer et al., 2011) | one year
  The HAPA variables include a stage assessment of behaviour change: Have you performed moderate physical for 30 minutes or longer on a minimum of 3 days per week? (rating: No, and I don't intend to do so - No, but I am currently thinking about that - No, but I strongly intend to do so - Yes, but it is difficult to me - Yes and it is easy to me) Further more, the HAPA variables include a validation item ("Since when are you regularly active as you are now?") and sets of items about the participants' intention, self-efficacy, action and coping planning, risk perception, expectations of consequences of physical activity behaviour and action control regarding physical activity. See Schwarzer et al., 2011 (Rehabilitation psychology 56(3), 161-170) for more details. Furthermore, experiences with physical activity are included (Fleig et al., 2011).
Health-related Quality of Life (SF-12) (Bullinger, Kirchberger, 1998) | one year
Depression (PHQ-D) (Löwe et al., 2002) | one year
Perceived Stress scale (Cohen, Williamson, 1988) | one year
Attitudes towards performing sports (Brand, 2006) | one year
  Four items assess the attitudes towards performing physical activity which are based on cognitions (e.g. "When I think about it, I regard physical activity as: not healthy -- very healthy"). Four items assess the attitudes based on affective judgement (e.g. "When I think about bein physically active, I feel not satisfied -- very satisfied"). Each of the eight items is rated on a 7-point scale in between the two poles.
Questionnaire for the detection of pain coping strategies (FESV) (Geissner, 2001) | one year
Tampa Scale of Kinesiophobia (TSK) (Kori et al., 1990) | one year
Avoidance-Endurance Questionnaire (AEQ) (Hasenbring et al., 2009) | one year

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Institute of Sport Science and Sport, Erlangen, Bavaria
  - Paracelsus-Klinik an der Gande, Bad Gandersheim, Lower Saxony
  - Klinik Weser, Bad Pyrmont, Lower Saxony

REFERENCES:
- [Background] Hofmann J, Peters S, Geidl W, Hentschke C, Pfeifer K. Effects of behavioural exercise therapy on the effectiveness of a multidisciplinary rehabilitation for chronic non-specific low back pain: study protocol for a randomised controlled trial. BMC Musculoskelet Disord. 2013 Mar 11;14:89. doi: 10.1186/1471-2474-14-89. PMID 23496822
- [Derived] Semrau J, Hentschke C, Peters S, Pfeifer K. Effects of behavioural exercise therapy on the effectiveness of multidisciplinary rehabilitation for chronic non-specific low back pain: a randomised controlled trial. BMC Musculoskelet Disord. 2021 May 29;22(1):500. doi: 10.1186/s12891-021-04353-y. PMID 34051780
- See also: Homepage: Research funding for care-oriented research "Chronic diseases and patient orientation" — http://www.forschung-patientenorientierung.de/index.php/projekte/zweite-foerderphase/modul-zwei-phase-2/vmo-vbt-pfeifer.html